CLINICAL TRIAL: NCT06531018
Title: Efficacy of Eltrombopag & Prednisolone Versus Prednisolone Monotherapy in Newly Diagnosed Immune Thrombocytopenia- A Randomized Control Trial
Brief Title: Role of Eltrombopag as First Line Therapy in Primary Immune Thrombocytopenia.
Acronym: EIT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renata PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 55603092023
Record Dates: First submitted 2024-07-06; First posted 2024-07-31 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: Primary ITP; Eltrombopag; First-line Therapy
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eltrombopag Arm (Experimental): Eltrombopag + Prednsolone
  Interventions: Drug: Eltrombopag 25 MG; Drug: Prednisolone
- Prednisolone alone arm (Placebo Comparator): Placebo + Prednisolone
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Eltrombopag 25 MG — Eltrombopag 25 mg daily and Prednisolone 1-2mg/kg, selected by block randomization from Day1 to Day 28. Both investigators and patients will be blinded.
  Other Names: Prednisolone
  Arms: Eltrombopag Arm
Drug: Prednisolone — Prednisolone 1-2 mg/kg and Placebo(same as eltrombopag 25mg Tablet), selected by block randomization from Day1 to Day 28. Both investigators and patients will be blinded.
  Other Names: Placebo

SUMMARY:
This will be a double-blind, placebo-control, randomized clinical trial conducted in the Department of Hematology, DMCH for one year. This study will help to establish the role of eltrombopag as a first-line therapy in newly diagnosed ITP. Newly diagnosed ITP patients will be selected after meeting inclusion and exclusion criteria, they will be thoroughly informed about the study, used drugs, randomization, risks, benefits, and follow-up. If they agree to participate, their consent will be taken and they will be enrolled in the study. A detailed history and clinical exam will be done. Primary investigation will be - CBC PBF, RBS, ANA, TSH, Anti H. pyloriIgG, Anti-HCV, APTT, and BMS (if indicated). The main outcome variable will be platelet count and number of spontaneous bleeding. Total sample size would be 100 (50 in each group). Enrolled patients would be divided into two groups (1:1) by block randomization. One group will get Eltrombopag& Prednisolone and other group will get Eltrombopag& Placebo. Researchers or any one related to the study in DMCH, patients & their attendants, no one will know which patient will get placebo or eltrombopag. Only a respectable third party will know the information. A patient would be followed up on 1st, 2nd and 4th week of starting therapy. Patients would be evaluated in every follow up by history, physical examination and investigation. History of any spontaneous bleeding event, any discomfort or new symptoms science last follow up will be noted. General examination will be performed in every follow-up. CBC, RBS, ALT, AST, creatinine will be done in every follow-up. Data will be collected on a pre-designed case record form and will be collected through face-to-face interviews, physical examination, and laboratory reports. After data collection data will be edited, cleaned, and prepared for analysis at the end of the study. The statistical analysis will be conducted using SPSS version 25 statistical software. The results of the study will be published in national and international journals.

DETAILED DESCRIPTION:
Study procedure After meeting inclusion and exclusion criteria patients will be thoroughly informed about the study, used drugs, randomization, risk and benefits, follow up. If they agree to participate in the study, their consent for this study will be taken and they will be enrolled in the study.

Detail history and clinical exam will be done. Key points are- History of spontaneous bleeding in last month, History of vaccination, History of recent viral infection, fever, Presence of organomegaly.

Primary investigation will be- CBC PBF, RBS, ANA, TSH, Anti H. pyloriIgG, Anti-HCV, APTT, BMS (if indicated)

NB:

1. If APTT is more than 10 sec of control, patient would be evaluated for Anti-Phospholipid Syndrome by anti-cardiolipin Antibody and Anti-beta2 glycoprotein1 Antibody
2. If Hemoglobin in less than 11.5gm/dL patient would be evaluated for Anemia by Iron Profile or Coomb's Test based on CBC parameter and PBF findings] Randomization: Enrolled patients would be divided into two groups (1:1) by block randomization. Block Randomization would be done by computer generated pattern. Actual randomization plan will be provided by Renata limited team who know about eltrombopag and placebo. Randomization allocation delivered only to the enrolling site study staff. A voluntary nurse will be in charge of enrolling the patients according to randomization plan.

Blinding and placebo control: It will be a double-blind study. Researchers nor participants will know who is getting placebo/eltromopag. One group will get Prednisolone & Eltrombopag and another group will get Prednisolone & Placebo. Eltrombopag, Prednisolone and Placebo will be provided by Renata Limited Bangladesh and patient will get at free of costs. Placebo will have same size, shape, color, markings, taste, smell and packaging like Eltrombopag. Eltrombopag and placebo will be provided in separate color-coded box marked-A (red) or B (green). Group A and Group B participants will be given colored cards (red and green) for identification. They will receive tablets from marked box. Researchers or any one related to the study in DMCH, patients & their attendants no will know which box contain placebo or eltrombopag. Only respectable person of Renata limited will know the information. The team who knows the information will be head by their CEO. At the end point all data will be submitted to the team who know about placebo.

Experimental Group - Eltrombopag& Prednisolone Control Group - Prednisolone and Placebo Dose- Prednisolone 1mg/kg/day for 28 days Eltrombopag/Placebo 25mg/day for 28 days Follow Up- Follow up at the end of 1st week, 2nd week and 4th week Patient would be evaluated in every follow up by history, physical examination and investigation. History of any spontaneous bleeding event, any discomfort or new symptoms science last follow up. General examination will be performed in every follow up. CBC, RBS, ALT, AST and creatinine will be done in every follow up.

Primary End Point-28 days after starting therapy. Complete Response is expected after 28 days of therapy.

Patient would continue therapy and follow up in OPD but would not be included in the study.

Supportive care and rescue- A Data and Safety Monitoring Board (DSMB) will be formed which will include two members of NREC, one hematologist and one medicine specialist. Any adverse event (Drugs side effects- headache, weight gain, changes in liver enzymes, high blood sugar) or serious adverse event (grade 3 or grade 4 bleeding, hospitalization, thrombosis) will be delt with proper medical care.

If any patient shows no response within 14 days and has grade 3 or 4 bleeding rescue with methyl prednisolone or IV Ig would be given and discontinued from study. If group A patient reaches platelet count >400x109\L, eltrombopag will be stopped.

Data Analysis After data collection data will be edited, cleaned and prepared for analysis at the end of the study. At the end of the study, all data will be submitted to the team who know about placebo/eltrombopag. The statistical analysis will be conducted using SPSS (statistical package for the social science) version 25 statistical software. The findings of the study will be presented by frequency and percentage in tables. Means and standard deviations for continuous variables and proportion for categorical variables will be used to describe the characteristics of the total sample. Association between two qualitative variables will be assessed by Chi-square test, where p<0.05 with 95% confidence level will be considered as significant. Appropriate statistical tests will be done to interpret the findings of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed ITP
2. Platelet Count ≤ 30x109/L
3. Age between 18 to 70 years.

Exclusion Criteria:

1. Persistent or chronic ITP
2. Pregnant women
3. Secondary ITP- ITP due to SLE, Anti-phospholipid syndrome, Evans syndrome, HCV or H Pylori associated ITP.
4. History of vaccination, recent viral infection, fever
5. Evan's Syndrome
6. Known case of chronic renal failure or liver diseases
7. Grade 3 or 4 bleeding at presentation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Platelet count | 28 days (platelet count will be measured at the end of 1st, 2nd and 4th week)
  Compare change in platelet count in two groups
Spontaneous bleeding | 28 days (Spontaneous bleeding episodes will be noted by face to face interview at the end of 1st, 2nd and 4th week)
  Compare number of Spontaneous bleeding in two groups

SECONDARY OUTCOMES:
Changes in hemoglobin | 28 days (hemoglobin will be measured at the end of 1st, 2nd and 4th week)
  Compare change in hemoglobin count in two groups
Changes in Total WBC count | 28days (WBC count will be measured at the end of 1st, 2nd and 4th week)
  Compare change in total WBC count in two groups
Change in ALT | 28 days ( ALT will be measured at the end of 1st, 2nd and 4th week)
  Compare change in ALT in two groups
Change in AST | 28 days ( AST will be measured at the end of 1st, 2nd and 4th week)
  Compare change in AST
Change in S.Createnine | 28 days (S.Createnine will be measured at the end of 1st, 2nd and 4th week)
  Compare change in S.Createnine in two groups
Change in RBS | 28 days (RBS will be measured at the end of 1st, 2nd and 4th week)
  Compare change RBS in two groups

CONTACTS AND LOCATIONS:
Overall Officials: Md Manirul Islam, MBBS,FCPS, Principal Investigator — Dhaka Medical College
Locations (1):
- Dhaka Medical College Hospital, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Sharing via E-Mail of PI and will be also available in DMC database.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From the starting of data collection to upto one year of the end of the study.
Access Criteria: Via submitting request to PI via EMail

REFERENCES:
- [Result] Gomez-Almaguer D, Herrera-Rojas MA, Jaime-Perez JC, Gomez-De Leon A, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Tarin-Arzaga L, Hernandez-Reyes J, Ruiz-Arguelles GJ. Eltrombopag and high-dose dexamethasone as frontline treatment of newly diagnosed immune thrombocytopenia in adults. Blood. 2014 Jun 19;123(25):3906-8. doi: 10.1182/blood-2014-01-549360. Epub 2014 May 6. PMID 24802773
- [Result] Gomez-Almaguer D, Colunga-Pedraza PR, Gomez-De Leon A, Gutierrez-Aguirre CH, Cantu-Rodriguez OG, Jaime-Perez JC. Eltrombopag, low-dose rituximab, and dexamethasone combination as frontline treatment of newly diagnosed immune thrombocytopaenia. Br J Haematol. 2019 Jan;184(2):288-290. doi: 10.1111/bjh.15070. Epub 2017 Dec 21. No abstract available. PMID 29270980
- [Result] Gomez-Almaguer D. Eltrombopag-based combination treatment for immune thrombocytopenia. Ther Adv Hematol. 2018 Oct 4;9(10):309-317. doi: 10.1177/2040620718798798. eCollection 2018 Oct. PMID 30344993
- [Result] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Result] Shimano KA, Grace RF, Despotovic JM, Neufeld EJ, Klaassen RJ, Bennett CM, Ma C, London WB, Neunert C. Phase 3 randomised trial of eltrombopag versus standard first-line pharmacological management for newly diagnosed immune thrombocytopaenia (ITP) in children: study protocol. BMJ Open. 2021 Aug 27;11(8):e044885. doi: 10.1136/bmjopen-2020-044885. PMID 34452956

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT06531018/Prot_SAP_ICF_000.pdf